CLINICAL TRIAL: NCT00266838
Title: A Double Blind Interventional Study of the Efficacy of Topical Eye Treatment in the Prevention of Docetaxel Induced Dacryostenosis
Brief Title: Prevention of Docetaxel Induced Dacryostenosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Ilse Mombaerts, UZLeuven
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UZL OFT-ML 3386
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2005-12

CONDITIONS: Epiphora
Keywords: Lacrimal Obstruction; Epiphora
MeSH Terms: conditions — Lacrimal Apparatus Diseases | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lacrystat (Placebo Comparator): Lacrystat
  Interventions: Drug: Maxidex; Lacrystat
- Maxidex (Active Comparator): Applying Maxidex
  Interventions: Drug: Maxidex; Lacrystat

INTERVENTIONS:
Drug: Maxidex; Lacrystat — 6 times daily, for 20 weeks.

SUMMARY:
The antineoplastic agent Docetaxel (Taxotere®) is approved for the treatment of patients with metastatic and locally advanced breast cancer and other malignancies. There are 2 frequently used schedules of treatment with Docetaxel. Docetaxel can be administered every 3 weeks or in a weekly regimen. The efficacy seems to be similar but the toxicity profile changes. In the standard 3-weekly Docetaxel regimen the dose-limiting side effect is myelosuppression, while in the weekly regimen there is only a mild myelosuppression. On the other hand, weekly Docetaxel has a side effect that is rare in the 3-weekly schedule: epiphora (= tearing eye) caused by dacryostenosis.

The underlying mechanism of dacryostenosis induced by weekly Docetaxel is fibrosis of the lacrimal puncta and canaliculi. Docetaxel has been reported to be secreted in the lacrimal tears. Direct contact between Docetaxel containing tears and the epithelial lining causes chronic inflammation of the mucosa and ultimately fibrosis of the most narrow part of the lacrimal outflow system i.e. the lacrimal puncta and canaliculi.

A surgical treatment is possible for dacryostenosis. In case of subtotal stenosis of the lacrimal canaliculi, silicone intubation of the canaliculi is performed in order to prevent further closure. In the case of complete stenosis, placement of a permanent pyrex glass tube of Jones is required.

To our knowledge, there is no primary prevention for Docetaxel induced dacryostenosis.

The rationale of this randomized double blind interventional study is to investigate the efficacy of corticosteroid versus artificial tears topical eye treatment in patients on a weekly Docetaxel regimen in prevention of dacryostenosis. The dacryotoxic agent Docetaxel in the lacrimal tears will be washed away by the repetitive use of eye drops. In addition, eye drops containing corticosteroids have an anti-inflammatory effect and may further prevent the formation of fibrosis.

A new treatment protocol will be investigated. Two different commercially available eye drops will be compared: dexamethasone sodium phosphate (Maxidex®, Alcon) in one eye of the patient and artificial tears (Lacrystat®, Viatris) in the other eye of the same patient. The study period will start with topical eye treatment from day 1 of cycle 1 and will continue during the administration of chemotherapy, with a final analysis at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic breast cancer receiving weekly Docetaxel chemotherapy with rest weeks in between at regular time intervals. The timing of rest weeks between cycles is not restricted. Examples of allowed regimens are Docetaxel 36 mg/m2 day 1 and 8 every 3 weeks; day 1, 8, 15 every 4 weeks; day 1, 8, 15, 21, 28, 35, 42, 49 every 10 weeks. Dosing and rest weeks can be further modified depending on the clinical situation, but dose intensity should be at least 60 mg/m2 every 3 weeks during the 9 week treatments for eligibility. Combination with other chemotherapy (such as capecitabine) is allowed.
* Capability to administer eye drops (either by patient or companion).
* Written informed consent.
* Age > 18 y

Exclusion Criteria:

* Systemic criteria:

  * Previous administration of Docetaxel.
  * Pregnancy.
* Eye criteria:

  * Ocular surface, corneal, conjunctival or eyelid disease.
  * Soft contact lens wearing
  * Glaucoma
* Lacrimal criteria:

  * Hypersecretion of tears: ocular surface, corneal, conjunctival or eyelid disease.
  * Functional blockage of lacrimal drainage without anatomical obstruction (facial nerve palsy, displacement of the lower lacrimal punctum from the lacrimal lake, involutional lower eyelid laxity).
  * Anatomical obstruction of lacrimal drainage system:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of dacryostenosis | 20 weeks
Grading of dacryostenosis | 20 weeks

SECONDARY OUTCOMES:
Correlation Docetaxel in lacrimal tear and dacryostenosis | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Mombaerts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Mombaerts, Leuven, Belgium